CLINICAL TRIAL: NCT01704859
Title: VITamin D and OmegA-3 TriaL (VITAL): Fractures, Vitamin D and Genetic Markers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Meryl LeBoff, Director of Skeletal Health and Osteoporosis Center, Brigham and Women's Hospital
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: 2010P002005; 1R01AR070854-01A1 (NIH)
Record Dates: First submitted 2012-10-09; First posted 2012-10-12 (Estimated); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Fractures
Keywords: fracture
MeSH Terms: conditions — Fractures, Bone | interventions — Fatty Acids, Omega-3; Fish Oils; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Vitamin D placebo + fish oil placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Vitamin D3 placebo; Dietary Supplement: Fish oil placebo
- Vitamin D placebo + fish oil (Active Comparator)
  Interventions: Dietary Supplement: Vitamin D3 placebo; Drug: omega-3 fatty acids (fish oil)
- Vitamin D + fish oil placebo (Active Comparator)
  Interventions: Dietary Supplement: Fish oil placebo; Dietary Supplement: Vitamin D3
- Vitamin D + fish oil (Active Comparator)
  Interventions: Drug: omega-3 fatty acids (fish oil); Dietary Supplement: Vitamin D3

INTERVENTIONS:
Dietary Supplement: Vitamin D3 placebo — Vitamin D placebo
  Arms: Vitamin D placebo + fish oil; Vitamin D placebo + fish oil placebo
Dietary Supplement: Fish oil placebo — Fish oil placebo
  Arms: Vitamin D + fish oil placebo; Vitamin D placebo + fish oil placebo
Drug: omega-3 fatty acids (fish oil) — Omacor, 1 capsule per day. Each capsule of Omacor contains 840 milligrams of marine omega-3 fatty acids (465 mg of eicosapentaenoic acid [EPA] and 375 mg of docosahexaenoic acid [DHA]).
  Arms: Vitamin D + fish oil; Vitamin D placebo + fish oil
Dietary Supplement: Vitamin D3 — Vitamin D3 (cholecalciferol), 2000 IU per day.
  Other Names: cholecalciferol
  Arms: Vitamin D + fish oil; Vitamin D + fish oil placebo

SUMMARY:
The VITamin D and OmegA-3 TriaL (VITAL; NCT 01169259) is a randomized clinical trial in 25,871 U.S. men and women investigating whether taking daily dietary supplements of vitamin D3 (2000 IU) or omega-3 fatty acids (Omacor® fish oil, 1 gram) reduces the risk of developing cancer, heart disease, and stroke in people who do not have a prior history of these illnesses. This ancillary study is being conducted among participants in VITAL and will examine (1) whether vitamin D reduces incident total, non-vertebral fractures, and hip fractures and (2) whether this reduction is modified by vitamin D levels

DETAILED DESCRIPTION:
The VITAL: Vitamin D, Fractures, and Genetic Markers is an ancillary study of the parent VITAL trial (VITamin D and OmegA-3 TriaL). The study will require the adjudication of all self-reported incident fracture events among 25,871 men and women. Findings from this ancillary study will inform clinical practice on the role(s) of vitamin D supplements in fracture prevention. This proposal will generate important positive or informative negative results about effects of supplemental vitamin D3 alone on fracture risk, while also elucidating the relative importance of vitamin D biomarkers and genetic variations in vitamin D-related pathways on bone. Findings from the proposed ancillary study have the potential for major clinical as well as public health impact for both men and women in the U.S.

ELIGIBILITY:
All participants from the VITAL parent study (NCT01169259) were enrolled in this ancillary study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25871 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-11-23 (Actual)

PRIMARY OUTCOMES:
Incident total, non-vertebral, and hip fractures | 5 years
  To determine whether vitamin D supplementation will reduce incident total, non-vertebral, and hip fractures according to annual questionnaires, medical record review, and fracture adjudication.

SECONDARY OUTCOMES:
Incident total, non-vertebral, and hip fractures | 5 years
  To determine whether baseline vitamin D levels and genetic variation in vitamin D-related pathways modify effects of vitamin D supplements on fractures.

CONTACTS AND LOCATIONS:
Overall Officials: Meryl S LeBoff, M.D., Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] LeBoff MS, Yue AY, Copeland T, Cook NR, Buring JE, Manson JE. VITAL-Bone Health: rationale and design of two ancillary studies evaluating the effects of vitamin D and/or omega-3 fatty acid supplements on incident fractures and bone health outcomes in the VITamin D and OmegA-3 TriaL (VITAL). Contemp Clin Trials. 2015 Mar;41:259-68. doi: 10.1016/j.cct.2015.01.007. Epub 2015 Jan 24. PMID 25623291
- [Background] LeBoff MS, Chou SH, Murata EM, Donlon CM, Cook NR, Mora S, Lee IM, Kotler G, Bubes V, Buring JE, Manson JE. Effects of Supplemental Vitamin D on Bone Health Outcomes in Women and Men in the VITamin D and OmegA-3 TriaL (VITAL). J Bone Miner Res. 2020 May;35(5):883-893. doi: 10.1002/jbmr.3958. Epub 2020 Jan 30. PMID 31923341
- [Background] LeBoff MS, Chou SH, Ratliff KA, Cook NR, Khurana B, Kim E, Cawthon PM, Bauer DC, Black D, Gallagher JC, Lee IM, Buring JE, Manson JE. Supplemental Vitamin D and Incident Fractures in Midlife and Older Adults. N Engl J Med. 2022 Jul 28;387(4):299-309. doi: 10.1056/NEJMoa2202106. PMID 35939577
- [Derived] Chou SH, Murata EM, Yu C, Danik J, Kotler G, Cook NR, Bubes V, Mora S, Chandler PD, Tobias DK, Copeland T, Buring JE, Manson JE, LeBoff MS. Effects of Vitamin D3 Supplementation on Body Composition in the VITamin D and OmegA-3 TriaL (VITAL). J Clin Endocrinol Metab. 2021 Apr 23;106(5):1377-1388. doi: 10.1210/clinem/dgaa981. PMID 33513226
- [Derived] LeBoff MS, Murata EM, Cook NR, Cawthon P, Chou SH, Kotler G, Bubes V, Buring JE, Manson JE. VITamin D and OmegA-3 TriaL (VITAL): Effects of Vitamin D Supplements on Risk of Falls in the US Population. J Clin Endocrinol Metab. 2020 Sep 1;105(9):2929-38. doi: 10.1210/clinem/dgaa311. PMID 32492153
- See also: VITAL study website — http://www.vitalstudy.org/